CLINICAL TRIAL: NCT05285891
Title: Randomized, Blinded Discontinuation Trial of Ocrelizumab in Early Relapsing Multiple Sclerosis (AMS05)
Brief Title: Ocrelizumab Discontinuation in Relapsing Multiple Sclerosis
Acronym: AMS05
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (ACE) (Unknown); Rho Federal Systems Division, Inc. (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT AMS05
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Ocrelizumab; Multiple sclerosis; Relapse
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ocrelizumab Arm (Experimental): All eligible participants will be initiated on OCR using the standard approved administration schedule of two 300 mg infusions separated by 14 days (i.e., Days 0 and 14) for a total of 600 mg, followed by 600 mg infusions at Month 6, 12, 18, and 24.
  In this arm participants will continue to receive OCR infusions every 6 months through Month 48.
  Interventions: Drug: Ocrelizumab
- Placebo Arm (Placebo Comparator): All eligible participants will be initiated on OCR using the standard approved administration schedule of two 300 mg infusions separated by 14 days (i.e., Days 0 and 14) for a total of 600 mg, followed by 600 mg infusions at Month 6, 12, 18, and 24.
  In this arm, starting at Month 30, participants will receive placebo infusions every 6 months through Month 48.
  Interventions: Drug: Placebo for Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Two 300 mg intravenous (IV) OCR infusions separated by 14 days (i.e., Days 0 and 14) for a total of 600 mg, followed by 600 mg OCR infusions every 6 months from Month 6 through Month 48.
  Other Names: Ocrevus
  Arms: Ocrelizumab Arm
Drug: Placebo for Ocrelizumab — Placebo infusions every 6 months from Month 30 through Month 48.
  Arms: Placebo Arm

SUMMARY:
This study is a prospective, multi-center, randomized, double blinded, placebo-controlled study of OCR treatment-discontinuation in patients with early RMS. All eligible participants will be initiated on OCR using the standard approved administration schedule of two 300 mg infusions separated by 14 days (i.e., Days 0 and 14) for a total of 600 mg, followed by 600 mg infusions at Month 6,12, 18, and 24. At Month 24, participants will be randomized (2:1) to one of two Arms with randomized treatment beginning at Month 30: Arm 1: placebo infusions every 6 months; or Arm 2: OCR infusions every 6 months. The treatment period will be for a total of 48 months.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized, double blinded, placebo-controlled study of OCR treatment-discontinuation in patients with early RMS. All eligible participants will be initiated on OCR using the standard approved administration schedule of two 300 mg infusions separated by 14 days (i.e., Days 0 and 14) for a total of 600 mg, followed by 600 mg infusions at Month 6, 12, 18, and 24. At Month 24, participants will be randomized (2:1) to one of two Arms with randomized treatment beginning at Month 30: Arm 1: placebo infusions every 6 months; Arm 2: OCR infusions every 6 months. The treatment period will be for a total of 48 months.

The study will consist of the following periods, with participants undergoing study assessments, including physical exams, neurological exams, EDSS, LCLA, SDMT, MFIS, MSQOL-54, PHQ9, EQ-5D-5L, and frequent co-registered research-quality MRI to sensitively assess for new inflammatory disease activity (new or enlarging T2 lesions), under schedules described in detail below. Biological sampling includes blood samples for functional immune profiling and stool samples for microbiome studies. Biomarker-based assessments are to include but not be limited to NfL and B cell levels.

Screening Period:

After obtaining informed consent, all screening assessments, and procedures to establish eligibility will be performed. These may be completed during one or more study visits within the 30-day screening window. Biological sampling with associated MRIs will include 2 samples obtained prior to initiation of OCR treatment.

Open-label Treatment Period:

Participants that meet all eligibility criteria for enrollment will be initiated on OCR using the standard approved administration and will be followed for 24 months under the standard of care clinical efficacy and safety monitoring described below. Biological sampling occurs at 6, 12, 18, and 24 months as well as prior to the 12 and 24 months visits (14 days +/- 7 days of the visit). MRIs will occur at 6, 12, 18, and 24 months.Participants who discontinue study therapy during the open-label treatment period are asked to return for an early withdrawal visit and a safety follow-up phone call approximately 6 months after their last dose.

Blinded Treatment Period:

At Month 24, participants will be randomized (2:1) to either: (Arm 1) placebo infusions every 6 months; or (Arm 2) continue with OCR infusions every 6 months. The blinded treatment period will extend to Month 48 or until new disease activity is observed. All participants in the blinded treatment period will be closely monitored clinically and with frequent research MRIs using a standard protocol that assesses for the development of any new inflammatory disease activity observed following Month 24. The development of such new inflammatory disease activity will represent the primary study endpoint. It will be defined as one or more of the following: (1) one or more new clinical relapse(s) (see relapse definition in section 3.2) or (2) MRI evidence on frequent (every 3 months) serial scans of new disease activity. The central imaging analysis will identify incident new or enlarging MRI T2 lesions as compared to prevalent brain lesions documented in each participant from Month 24 and thereafter.

Frequent biological sampling will include blood samples collected every 3 months and stool samples collected every 6 months through the 48-month end of study.

Unblinded Follow-up period:

For participants who discontinue blinded study therapy before Month 48, including those meeting the primary endpoint by manifesting new disease activity following Month 24 as defined above, blinded treatment allocation will be revealed and discussed, as described in section 3.5.1. Participants may choose to receive OCR or other treatment and are encouraged to continue with study assessments per the schedule of events. For participants that meet the primary endpoint, OCR will be provided by the study for those who choose to receive OCR after unblinding and continue with study assessments per the schedule of events.

Functional immune response profiles of reconstituting B cells as well as non-B cells (T cells and myeloid cells) will be compared between participants who do, versus those do not, benefit from durable remission of relapsing biology, to identify cellular immune response profiles that may underlie the state of durable tolerance versus lack of durable tolerance.

Safety Follow-up:

Participants who are treated with OCR through Month 48 will have a phone visit 6 months after their last dose. If there are safety concerns, the participant can be brought in for an unscheduled visit.

ELIGIBILITY:
Inclusion Criteria:

1. Have at least one clinical episode that satisfies McDonald 2017 criteria for early Multiple sclerosis (MS) with a dissemination in time that can be met clinically, by Magnetic Resonance Imaging (MRI), or based on oligoclonal band (OCB) positivity
2. Have a length of disease duration, from first symptom, of ≤ 3 years at time of informed consent
3. For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use effective methods of contraception during the treatment period and for at least 6 months after the last dose of study drug:

   1. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
   2. Examples of contraceptive methods include bilateral tubal ligation, male sterilization, established hormonal contraceptives that inhibit ovulation, hormone- releasing intrauterine devices, and copper intrauterine devices
   3. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception
   4. Barrier methods must always be supplemented with the use of a spermicide

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol
2. History of primary progressive multiple sclerosis (PPMS), progressive relapsing multiple sclerosis (PRMS), or secondary progressive multiple sclerosis (SPMS)
3. Any metallic material or electronic device in the body, or condition that precludes the participant from undergoing MRI
4. Known presence or history of other neurological disorders, including but not limited to the following:

   * Ischemic cerebrovascular disorders, including but not limited to transient ischemic attack, subarachnoid hemorrhage, cerebral thrombosis, cerebral embolism, or cerebral hemorrhage
   * CNS or spinal cord tumor, metabolic or infectious cause of myelopathy, genetically inherited progressive CNS disorder, CNS sarcoidosis, or systemic autoimmune disorders potentially causing progressive neurologic disease or affecting ability to perform the study assessments
5. Pregnancy or lactation

   • Female participants of childbearing potential must have a negative urine pregnancy test at screening
6. Any concomitant disease that may require chronic systemic treatment with corticosteroids or immunosuppressants during the course of the study
7. Lack of peripheral venous access
8. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
9. Significant, inadequately controlled (e.g., diagnostic evaluations indicated or change in medications warranted) disease, such as cardiovascular (including cardiac arrhythmia), pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine, and gastrointestinal or any other significant disease that in the opinion of the investigator may preclude participant from participating in the study
10. Functional status of New York Heart Association (NYHA) Class III or higher for heart failure at the screening visit
11. Known active bacterial, viral, fungal, mycobacterial infection or other infection (including tuberculosis (TB) or atypical mycobacterial disease but excluding limited superficial fungal or viral infections of the skin or nails) or any severe episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks prior to Mo 0/Day 0 infusion or oral antibiotics within 2 weeks prior to Mo 0/Day 0 infusion
12. Active or chronic infection with human immunodeficiency virus (HIV), syphilis or TB (see laboratory tests below)
13. Evidence of past hepatitis B (including treated hepatitis B) or untreated hepatitis C infection (treated hepatitis C is not considered exclusionary). Hepatitis B surface antibody following hepatitis B immunization is not considered to be evidence of past infection (see laboratory tests below).
14. Known active malignancy or active monitoring for recurrence of malignancy, including solid tumors and hematological malignancies, except basal cell, in situ squamous cell carcinoma of the skin, and in situ carcinoma of the cervix or the uterus that have been excised with clear margins
15. Substance use disorder, including the recurrent use of alcohol and/or drugs within the past year associated with clinically significant impairment associated with failure to meet major responsibilities at work, school, or home
16. Receipt of live or live-attenuated vaccines within 4 weeks prior to Mo 0/Day 0 infusion
17. Contraindications to or severe intolerance of oral or IV corticosteroids, including IV methylprednisolone administered according to the country label, including:

    * Psychosis not controlled by a treatment
    * Hypersensitivity to any of the constituents or excipients of the preceding steroids
18. Current or prior treatment with the following MS DMTs: fingolimod and other S1P receptor modulators, cladribine, natalizumab, anti-CD20 molecules, alemtuzumab, and chemotherapeutic agents
19. Treatment with fumarates within 30 days prior to collection of Mo 0/Day 0 mechanistic samples, Mo 0/Day 0 MRI, and Mo 0/Day 0 infusion
20. (a) Current or prior treatment with any approved or experimental immunomodulatory therapies, unless reviewed and approved by the SAC (Section 3.6), or (b) Treatment with any experimental procedure for MS (e.g., treatment for chronic cerebrospinal venous insufficiency)
21. Systemic corticosteroid therapy within 4 weeks prior to the collection of screening mechanistic samples and the screening MRI
22. Systemic corticosteroid therapy within 4 weeks prior to the Mo 0/Day 0 infusion
23. Screening laboratory test results as follows:

    * Positive infection screening tests for:

      i. Hepatitis B surface antigen (HbsAg) or hepatitis B core antibody (HbcAb) ii. Hepatitis C (HCV) antibody if positive screen for HCV RNA Polymerase Chain Reaction (PCR) iii. Rapid plasma reagin (RPR)
    * A reactive RPR test unless followed by a subsequent negative RPR OR
    * A reactive RPR test unless successful completion of treatment has been documented as well as a consultation with and clearance by infectious disease department iv. HIV v. At or within twelve months of screening:
    * Positive QuantiFERON®-TB Gold test or positive purified protein derivative tuberculin skin test (PPD) (>5mm induration, regardless of Bacille Calmette-Guerin (BCG) vaccine administration) unless completion of treatment has been documented for active TB OR
    * An indeterminate QuantiFERON®-TB Gold test unless followed by a subsequent negative PPD or negative QuantiFERON®-TB Gold test as well as a consultation with and clearance by infectious disease department
    * Levels of serum immunoglobulin G (IgG) < 3.3g/L
    * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.0 x the upper limit of normal (ULN)
    * Platelet count < 100,000 plt/µL (<100 x 10⁹/L)
    * Hemoglobin < 10 g/dL
    * Absolute neutrophil count < 1.5 x 10⁹/L
    * Absolute lymphocyte count < 1.2 x 10⁹/L
24. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Absence of clinical relapse | From Month 24 to Month 48
  Durable remission of relapsing disease activity.
  This is defined as the absence of new relapsing disease activity from Month 24 through Month 48. This includes absence of clinical relapse as well as absence of evidence of MS disease activity by MRI defined by new or enlarging T2 lesions.

SECONDARY OUTCOMES:
The change in Expanded Disability Status Scale (EDSS) score | Month 24 to Month 48
  The Expanded Disability Status Scale (EDSS) score has a minimal value of zero, and maximal value is 10, with higher scores meaning worse outcome.
Proportion of participants with a serious adverse event (SAE) | Month 0 to Month 48
Proportion of participants who experience at least one Grade 3 or higher adverse event | Month 0 to Month 48
  Using National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
  Adverse events will be graded on a scale from 1 to 5 according to the following standards in the NCI-CTCAE manual:
  Grade 1 = mild adverse event Grade 2 = moderate adverse event Grade 3 = severe or medically significant Grade 4 = life-threatening consequences; urgent intervention indicated Grade 5 = death
Proportion of participants with infections, Grade 3 or higher | Month 0 to Month 48
Proportion of participants with malignancies | Month 0 to Month 48
Proportion of participants experiencing infusion related reactions | Month 0 to Month 48
  Defined as any at least possibly related adverse reaction within 24 hours of infusion which are Grade 3 or higher events
The ratio of granulocyte-macrophage colony-stimulating factor (GM-CSF) expressing B-Cells to Interleukin 10 (IL-10) expressing B cells at Month 48 in participants who do versus do not exhibit durable disease remission | Month 24 to Month 48

CONTACTS AND LOCATIONS:
Overall Officials: Amit Bar-Or, M.D., Study Chair — University of Pennsylvania, Perelman School of Medicine: Department of Neurology
Locations (12):
- United States (12):
  - Yale School of Medicine, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - University of Pennsylvania, Perelman School of Medicine, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, McGovern Medical School, Houston, Texas
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access
URL: http://www.immport.org/home

REFERENCES:
- See also: Autoimmunity Centers of Excellence — https://www.autoimmunitycenters.org/
- See also: National Institute of Allergy and Infectious — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — https://www.niaid.nih.gov/about/dait